CLINICAL TRIAL: NCT05426356
Title: Sacral Fracture Fusion/Fixation for Rapid Rehabilitation
Acronym: SAFFRON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300900
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Fracture;Pelvis; Sacral Fracture; Sacroiliac; Fusion; Fragility Fracture; Insufficiency Fractures; Osteoporosis
Keywords: Elderly; Fragility fracture; Pelvic fracture fixation; SI Joint Fusion; Non-surgical management
MeSH Terms: conditions — Hip Fractures; Fractures, Stress; Osteoporosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to sacral fracture fixation and SI joint fusion using iFuse-TORQ vs. non-surgical management (NSM). There is a crossover component for subjects who fail NSM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-Surgical Treatment (Active Comparator): Non-surgical management (NSM) of sacral insufficiency or fragility fractures (SFIF)
  Interventions: Other: Non-Surgical Management
- Surgical Treatment (Experimental): Surgical fixation of sacral insufficiency or fragility fractures (SFIF) with concomitant fusion of the sacroiliac (SI) joint
  Interventions: Device: Surgical Intervention

INTERVENTIONS:
Device: Surgical Intervention — Surgical sacral fracture fixation and SI joint fusion using iFuse-TORQ
  Arms: Surgical Treatment
Other: Non-Surgical Management — Non-surgical management (NSM) is any treatment deemed appropriate for the subject that does not involve surgery.
  Arms: Non-Surgical Treatment

SUMMARY:
To determine the safety and efficacy of concomitant sacral fracture fixation and sacroiliac (SI) joint fusion vs. non-surgical management for patients with debilitating sacral fragility or insufficiency fractures

DETAILED DESCRIPTION:
SAFFRON is a prospective, multicenter, randomized, controlled trial of surgical fixation of sacral insufficiency or fragility fractures (SFIF) with concomitant fusion of the sacroiliac (SI) joint vs. nonsurgical management (NSM). The goal of the study is to demonstrate the safety, performance, effectiveness, and cost-effectiveness of use of iFuse-TORQ™ in the treatment of sacral fragility or insufficiency fractures vs. NSM.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 60 years of age at screening.
2. Posterior pelvic pain correlating with fracture location that began EITHER within 14 days of a low-energy traumatic event, OR in the last 60 days in the absence of a traumatic event
3. Imaging (X-ray, CT, or MRI) showing fracture of the sacrum (unilateral or bilateral)
4. Patient is either bedbound or must use a wheelchair to cover distances more than 50ft
5. Prior to fracture, patient was able to ambulate using a cane or unassisted
6. Medically stable to undergo either surgical or non-surgical treatment of index fracture.
7. Patient is willing and able to provide written informed consent
8. Patient is mentally able to comply with study protocol requirements

Exclusion Criteria:

1. Patient requires surgery to address fracture in the pelvic ring (NSM not feasible)
2. Anatomic anomalies/defects that would preclude safe and/or biomechanically acceptable placement of implants across the sacroiliac joint (SIJ) and into the sacrum
3. Sacral fracture potentially or definitely related to tumor
4. Any permanent implants already in the sacrum (including cement), ilium, or anterior pelvic ring that could interfere with placement of transiliac transsacral or iliosacral screws or iFuse-TORQ implants
5. History of recent (within 1 year) non-index pelvic fracture with nonunion of sacrum or ilium.
6. Other clinically active fragility fracture of spine, hip, arms, or legs that could impair recovery from sacral fracture
7. Uncontrolled psychiatric disease (e.g., dementia, schizophrenia, major depression, personality disorders) that could interfere with study participation or assessments
8. Prominent neurologic condition that would interfere with study participation including the use of electronic diaries (e.g., dementia) or recovery of mobility (e.g., severe diabetic neuropathy, multiple sclerosis)
9. Known allergy to titanium or titanium alloys
10. Current local or systemic infection that raises the risk of surgery.
11. Known or suspected active drug or alcohol abuse, including opioids.
12. Patient lives or plans to move more than 100 miles from the site during the course of the study.
13. Current enrollment in another investigational clinical trial related to fractures or osteoporosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Time following treatment initiation to reach a 2-point improvement in mobility from baseline as measured using self-rated Modified Functional Mobility scale (MFMS). | 1 year
  The study's primary efficacy endpoint is the time required to achieve an improvement from baseline (study entry) of 2 or more points on the Modified Functional Mobility scale. The scale is administered on a weekly basis following the initiation of treatment until achieving a 2-point improvement or the subject crosses over.
Proportion of subjects with serious adverse event (SAE) probably or definitely related to a complication of sacral fracture and/or associated treatment (both arms) or probably or definitely related to iFuse-TORQ (surgery only). | 1 year
  If randomized to surgery:
  Proportion of subjects with either:
  * Serious adverse event deemed probably or definitely related to iFuse-TORQ
  * Serious adverse event deemed probably or definitely a complication of sacral fracture and/or associated treatment
  If randomized to NSM:
  Proportion of subjects with:
  * Serious adverse event deemed probably or definitely a complication of sacral fracture and/or associated treatment

SECONDARY OUTCOMES:
Continuous Summary Physical Performance Score (CSPPS) | 1 year
  Change of CSPPS scores at 6 weeks and 12 months. Continuous Summary Physical Performance Score (CSPPS) is a scoring system based on the Short Physical Performance Battery (SPPB) that is optimized for use in the elderly.
Patient-Reported Outcomes Measurement Information System (PROMIS) physical function | 6 weeks
  Change from baseline in self reported PROMIS physical function score at 6 weeks. This domain is scored between 1 (unable to do) and 5 (can be done without difficulty).
Oswestry Disability Index | 6 weeks
  Change from baseline in self reported Oswestry Disability Index at 6 weeks. Calculated scores range from 0 (no disability) to 50 (completely disabled).
Numeric Rating Scale pain score | 6 weeks
  Change from baseline in self reported Numeric Rating Scale pain score at 6 weeks. Pain scale ranges from 0 (pain free) to 10 (max pain).

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Study Director — SI-BONE
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Bryan Health Medical Center, Lincoln, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Orthopedic Associates of Reading, Wyomissing, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia, Charlottesville, Virginia
  - Kadlec Clinic Northwest Orthopedic & Sports Medicine, Richland, Washington

IPD SHARING:
Plan to Share IPD: No